CLINICAL TRIAL: NCT04493567
Title: An Open-label, Randomized, Two-period Cross-over Study to Investigate the Relative Bioavailability of BMS-986036 in Healthy, Overweight, and Obese Participants Following Subcutaneous Administration Via Auto-injector Versus Pre-filled Syringe
Brief Title: Relative Levels of BMS-986036 in Blood Plasma in Healthy, Overweight, and Obese Participants Following Subcutaneous Administration Via Auto-injector Versus Pre-filled Syringe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MB130-101
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Pegbelfermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: 1 x BMS-986036 via auto-injector or pre-filled syringe (Experimental)
  Interventions: Drug: BMS-986036
- Part B: 2 x BMS-986036 via auto-injector or pre-filled syringe (Experimental)
  Interventions: Drug: BMS-986036

INTERVENTIONS:
Drug: BMS-986036 — Specified dose on specified days

SUMMARY:
The purpose of this study is to develop an auto-injector (AI) device for the BMS-986036 subcutaneous formulation that can be self-administered conveniently by participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy, overweight, obese, male and female participants, as determined by normal in medical history, physical examination (PE), electrocardiograms (ECGs), and clinical laboratory determinations
* Body mass index (BMI) of 25.0 kg/m2 to 40.0 kg/m2, inclusive i) Approximately 25% of participants will be overweight and have a BMI between 25 kg/m2 and 30 kg/m2, inclusive ii) Approximately 75% of participants will be obese and have a BMI > 30 kg/m2 to ≤ 40 kg/m2
* Women and men must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Inability to tolerate subcutaneous (SC) injections
* Inability to be venipunctured and/or tolerate venous access
* Any sound medical, psychiatric, and/or social reason as determined by the investigator

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 29 days
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to 29 days
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of C-terminal intact BMS-986036 | Up to 29 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 115 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 85 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 85 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 85 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 85 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 85 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 85 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 85 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 85 days
  The PR interval is the time from the onset of the P wave to the start of the QRS complex.
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS interval | Up to 85 days
  QRS interval: A combination of the Q wave, R wave and S wave, the "QRS complex" represents ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 85 days
  The QT interval on the ECG is measured from the beginning of the QRS complex to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF interval | Up to 85 days
  Corrected QT interval using Fridericia's formula (QTcF)
Incidence of clinically significant changes in physical examination findings | Up to 85 days
Number of participants with local injection site reactions | Up to 57 days
Number of participants with Antibodies to fibroblast growth factor 21 (FGF21) | Up to 57 days
Number of participants with Antibodies to BMS-986036 | Up to 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, Anaheim, California
  - ICON (LPRA) - Salt Lake, Salt Lake City, Utah

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm